CLINICAL TRIAL: NCT05610969
Title: To Serenade or To Sedate? That is Still The Question - A Followup Trial On Anxiolytic Options Before Peripheral Nerve Blocks
Brief Title: Music vs Midazolam During Preop Nerve Block Placement - Part 2 Study On Anxiolytic Options Before Peripheral Nerve Blocks
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: terminated due to lack of resources
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Veena Graff, Assistant Professor of Anesthesiology & Critical Care, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 842519
Record Dates: First submitted 2022-08-05; First posted 2022-11-09 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Nerve Block; Anxiety; Preoperative Anxiety
Keywords: Midazolam; Adjuvants, Anesthesia; Anti-Anxiety Agents; Hypnotics and Sedatives; Tranquilizing Agents; Anesthetics; GABA Modulators; GABA Agents; Central Nervous System Depressants; Physiological Effects of Drugs; Neurotransmitter Agents
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy; Midazolam

STUDY DESIGN:
Intervention Model Description: 1:1
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Music group (Active Comparator): self-selected music
  Interventions: Other: Music
- Midazolam group (Active Comparator): IV midazolam (1mg to 2mg max)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Other: Music — patients in this group will receive self-selected music after the golden moment has been completed between the patient, provider, and nursing staff
  Arms: Music group
Drug: Midazolam — patients in this group will receive IV midazolam (1mg to 2mg max) after the golden moment has been completed
  Other Names: Hypnovel; Versed
  Arms: Midazolam group

SUMMARY:
This study is evaluating music vs midazolam as a means of anxiolysis for preoperative single-shot nerve block placement.

DETAILED DESCRIPTION:
Preoperative anxiety is common and can adversely affect a patient's perioperative course by elevating stress markers, promoting fluctuations in hemodynamics and negatively impacting on postoperative recovery. Preoperative anxiety is routinely treated with pharmacologic agents such as midazolam, a benzodiazepine, which has known, undesirable side effects including respiratory depression, hemodynamic perturbations, and paradoxical effects such as hostility, aggression, and psychomotor agitation. The use of sedative medications requires continuous vital sign monitoring of patients by either anesthesia or nursing personnel and there is a question of whether midazolam helps reduce pre-procedural anxiety compared with placebo. Music is a non-pharmacologic intervention that has been shown to significantly decrease preoperative anxiety. This intervention can be used as an adjunct or even replace pharmacologic agents to help with preoperative anxiety. Music is a modality that is virtually harm-free and relatively cheap in cost. Patients who are unable to tolerate pharmacologic agents to treat preoperative anxiety can greatly benefit from non-pharmacologic options such as music.

Regional anesthesia procedures such as an ultrasound guided, peripheral nerve block is a common bedside procedure done preoperatively. Patients may have some anxiety prior to the administration of this nerve block procedure and may receive sedation for it. However, it is imperative not to over sedate them as constant feedback from the patient is necessary during the procedure. Commonly, midazolam is used to reduce this anxiety, but non-pharmacologic therapies can also reduce anxiety. In our recent published study, we evaluated the use of research-selected, relaxing music, to reduce anxiety before the nerve block is administered. In this study, we used noise-canceling headphones and played research-selected music as our anxiolytic music modality and compared this with midazolam. The findings showed no difference between both groups in the change in anxiety scores from after to before the nerve block, however patients had better satisfaction in the midazolam group and increased difficulty in communication in the music group. We attributed this to not allowing patients to choose their own selection of music and the use of noise-canceling headphones.

Therefore, in this follow-up study, we aim to evaluate the use of patient-selected music via non-noise canceling headphones as a preoperative anxiolytic prior to the administration of a bedside, peripheral nerve block procedure. This study will be conducted at an ambulatory surgical center in a university setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are >18 years of age
* Patients able to give informed consent in receiving a peripheral nerve block in the preoperative bay for their primary anesthetic and/or for their postoperative pain control

Exclusion Criteria:

* significant psychiatric disorder such as generalized anxiety disorder, panic disorder, depression, psychosis, bipolar disorder
* individuals who were incompetent to give informed consent
* pregnant and/or breast-feeding patients
* any underlying coagulopathy
* infection or other factors which would be a contraindication to receiving a peripheral nerve block
* hypersensitivity to midazolam
* history of renal impairment.
* Patients who were extremely anxious (scores greater than 50 on the State Trait Anxiety Inventory-6 (STAI-6) tool) were also excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veena Graff, MD, MS, Principal Investigator — University of Pennsylvania, Anesthesiology and Critical Care
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Music Group | Midazolam Group
Started | 15 | 21
Completed | 15 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Music Group | Midazolam Group | Total
Number analyzed (Participants) | 15 | 21 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 21 | 35
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (19.1) | 42 (18.1) | 42.3 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 14 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 11 | 15 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 21 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in STAI-6 Scores From Post to Pre
Description: Spielberger State-Trait Anxiety Inventory 6 Scale range is from 20 to 80. Higher the score, the higher the anxiety level is.
Time Frame: 1-2 minutes before conducting golden moment for nerve block placement and immediately after nerve block placement (less than 1 minute after)
Population: Due to lack of resources the study was terminated early and data collection is incomplete.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Group | Midazolam Group
Number analyzed (Participants) | 15 | 21
score on a scale
  Pre STAI-6: number analyzed (Participants) | 15 | 18
  Pre STAI-6 | 34 (7.02) | 35.17 (9.22)
  Post STAI-6: number analyzed (Participants) | 13 | 16
  Post STAI-6 | 28.19 (5.17) | 27.2 (5.00)

2. Secondary Outcome: Patient Satisfaction Scores of the Experience During Procedure
Description: Survey which assess satisfaction on a 10-point numeric rating scale Scale ranges from 0 to 10. A higher number indicates a higher satisfaction
Time Frame: immediately after nerve block placement (less than 1 minute after)
Population: Due to lack of resources the study was terminated early and data collection is incomplete.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Music Group | Midazolam Group
Number analyzed (Participants) | 15 | 21
units on a scale | 10 [8 to 10] | 9 [8 to 10]

3. Secondary Outcome: Provider Satisfaction Scores of the Experience During Procedure
Description: as for outcome 2
Time Frame: immediately after nerve block placement (less than 1 minute after)
Population: Due to lack of resources the study was terminated early and data collection is incomplete.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Music Group | Midazolam Group
Number analyzed (Participants) | 15 | 21
units on a scale | 10 [9 to 10] | 10 [8 to 10]

4. Secondary Outcome: Evaluation of Difficulties in Communication From Provider to Patient and Patient to Provider
Description: surveyed on a 5-point Likert scale Scale ranges from 1 to 5; the higher the number, the more difficult it is to communicate.
Time Frame: immediately after nerve block placement (less than 1 minute after)
Population: Due to lack of resources the study was terminated early and data collection is incomplete.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Music Group | Midazolam Group
Number analyzed (Participants) | 15 | 21
score on a scale
  Patient Perspective: number analyzed (Participants) | 14 | 21
  Patient Perspective | 1 [1 to 2] | 1 [1 to 2]
  Physician Perspective: number analyzed (Participants) | 15 | 20
  Physician Perspective | 1 [1 to 2] | 1 [1 to 2]

5. Secondary Outcome: Block Times - Time it Took to do the Block
Description: differences amongst music and midazolam group
Time Frame: start of doing the block to immediately after nerve block placement, less than 1 minute after
Population: Due to lack of resources the study was terminated early and data collection is incomplete.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Music Group | Midazolam Group
Number analyzed (Participants) | 13 | 21
minutes | 7 (2.03) | 7.95 (3.26)

ADVERSE EVENTS:
Time Frame: Adverse events were noted from the beginning of the block placement up to 30 minutes after end of block placement. Due to lack of resources the study was terminated early and data collection is incomplete.
Arm/Group | Music Group | Midazolam Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/21
Other Adverse Events (participants affected / at risk) | 0/15 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT05610969/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT05610969/ICF_001.pdf